

# **Trial Statistical Analysis Plan**

c20692486-01

| BI Trial No.: | 1361.3 |
|---|---|
| Title: | Bioequivalence of a fixed dose combination tablet of empagliflozin/linagliptin/metformin extended release compared to the free combination of empagliflozin, linagliptin, and metformin extended release tablets following oral administration in healthy male and female subjects (an open-label, randomised, single-dose, two-period, two-sequence crossover study) |
| Investigational Products: | Empagliflozin/linagliptin/metformin extended release fixed dose combination |
| Responsible trial statisticians: | |
| | Phone:<br>Fax: |
| | Phone:<br>Fax: |
| Date of statistical analysis plan: | 08 DEC 2017 SIGNED |
| Version: | FINAL |

Proprietary confidential information

© 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1361.3 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1. **TABLE OF CONTENTS**

| TITLE | PAGE | 1 |
|------------|------------------------------------------------|----|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | F TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 7 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | 8 |
| 5. | ENDPOINTS | |
| 5.1 | PRIMARY ENDPOINTS | |
| 5.2 | SECONDARY ENDPOINTS. | |
| 5.2.1 | Key secondary endpoints | |
| 5.2.2 | Secondary endpoints | |
| 5.3 | FURTHER ENDPOINTS | |
| 5.4 | OTHER VARIABLES | |
| 5.4.1 | Demographic and other baseline characteristics | |
| 6. | GENERAL ANALYSIS DEFINITIONS | 11 |
| 6.1 | TREATMENTS | |
| <b>6.2</b> | IMPORTANT PROTOCOL VIOLATION | |
| 6.3 | PATIENT SETS ANALYSED | 15 |
| 6.5 | POOLING OF CENTRES | 16 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | 16 |
| 7. | PLANNED ANALYSIS | |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | |
| 7.3 | TREATMENT COMPLIANCE | |
| 7.4 | PRIMARY ENDPOINTS | |
| 7.5 | SECONDARY ENDPOINTS | 21 |
| 7.5.1 | Key secondary endpoints | |
| 7.5.2 | Secondary endpoints | 21 |
| 7.7 | EXTENT OF EXPOSURE | 22 |
| <b>7.8</b> | SAFETY ANALYSIS | 22 |
| 7.8.1 | Adverse events | |
| 7.8.2 | Laboratory data | |
| 7.8.3 | Vital signs | |
| 7.8.4 | ECG | |
| 7.8.5 | Others | 25 |
| <b>Q</b> | REFERENCES | 26 |

| <b>Boehringer Ingelheim</b> |
|------------------------------|
| TSAP for BI Trial No: 1361.3 |

| Page | 3 | of | 28 |
|------|---|----|----|

| Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|

| 10 F | HSTORY | FABLE | 28 |
|------|--------|-------|----|

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1361.3 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES

| Table 6.1: 1 | Treatments and labels used in the analysis | 11 |
|--------------|--------------------------------------------|----|
| | Important protocol violations | |
| | Subject sets analysed | |
| | History table | |

TSAP for BI Trial No: 1361.3 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

| Term | Definition / description |
|---|---|
| ADS | Analysis dataset |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ANOVA | Analysis of variance |
| $AUC_{0	ext{-tz}}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
| AUC <sub>0-72</sub> | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 72 hours |
| $AUC_{0\infty}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity |
| BI | Boehringer Ingelheim |
| BWC | Bioavailability/Bioequivalence, within-subject design, time-controlled |
| CI | Confidence interval |
| $C_{max}$ | Maximum measured concentration of the analyte in plasma |
| CRF | Case report form |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CV | Arithmetic coefficient of variation |
| DBLM | Database lock meeting |
| DILI | Drug induced liver injury |
| ECG | Electrocardiogram |
| EudraCT | European Union Drug Regulating Authorities Clinical Trials |
| FDC | Fixed dose combination |
| gCV | Geometric coefficient of variation |
| gMean | Geometric mean |
| ICH | International Conference on Harmonisation |
| LLT | Lower level term |
| Max | Maximum |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Min | Minimum |

TSAP for BI Trial No: 1361.3 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|---|---|
| N | Number non-missing observations |
| O*C | Oracle Clinical |
| PK | Pharmacokinetics |
| PKS | PK parameter set |
| PT | Preferred term |
| PV | Protocol violation |
| qd | Quaque die (daily) |
| R | Reference treatment |
| RAGe | Report Appendix Generator system |
| REP | Residual effect period |
| RPM | Report planning meeting |
| $\mathrm{SAS}^{\circledR}$ | Statistical Analysis System |
| SD | Standard deviation |
| SOC | System organ class |
| T | Test treatment |
| t <sub>max</sub> | Time from dosing to maximum measured concentration of the analyte in plasma |
| TS | Treated set |
| TSAP | Trial statistical analysis plan |
| ULN | Upper limit of normal |
| WHO-DD | World Health Organization Drug Dictionary |
| XPKISTAT | Library of SAS® Macros for PK analysis |
| XR | Extended release |

#### 3. INTRODUCTION

As per ICH E9 (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This Trial statistical analysis plan (TSAP) assumes familiarity with the Clinical Trial Protocol (CTP). In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data will be stored in a trial database within the Oracle ClinicalTM (O\*C) system.

Pharmacokinetic (PK) parameters will be calculated using Phoenix WinNonlin<sup>TM</sup> software (version 6.3, Certara USA Inc., Princeton, NJ, USA).

The statistical analyses will be performed within the validated working environment CARE, including SASTM (current Version 9.4, by SAS Institute Inc., Cary, NC, USA), and a number of SASTM-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the CTR appendices).

## 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses as planned in the CTP will be performed and are described in more detail in this TSAP. The following change compared to the protocol will be made:

No 'Randomised set' will be defined in the TSAP as data of subjects randomised but discontinued before first administration of trial medication will not be entered in the case report form. A correct display of the 'Randomised set' would not be possible.

TSAP for BI Trial No: 1361.3

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5. ENDPOINTS

#### 5.1 PRIMARY ENDPOINTS

**Section 5.5.1.1 of the CTP:** *The following primary endpoints will be determined:* 

- $AUC_{0-tz}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) for empagliflozin and metformin
- $AUC_{0-72}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 72 h) for linagliptin
- $C_{max}$  (maximum measured concentration of the analyte in plasma) for empagliflozin, linagliptin, and metformin

#### 5.2 SECONDARY ENDPOINTS

#### 5.2.1 Key secondary endpoints

This section is not applicable as no key secondary endpoints have been defined in the CTP.

#### 5.2.2 Secondary endpoints

**Section 5.5.1.2 of the CTP:** *The following secondary endpoint will be evaluated for empagliflozin, linagliptin, and metformin:* 

•  $AUC_{0-\infty}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)

#### 5.3 FURTHER ENDPOINTS

### Pharmacokinetic (PK):

Pharmacokinetic parameters are further parameters of interest. For more detail see CTP Section 5.5.1.3.

#### Safety:

**Section 5.2.1 of the CTP:** *Safety and tolerability of the investigational drugs will be assessed based on:* 

- Adverse events (including clinically relevant findings from the physical examination)
- Safety laboratory tests
- 12-lead ECG

• *Vital signs (blood pressure, pulse rate)* 

#### 5.4 OTHER VARIABLES

# 5.4.1 Demographic and other baseline characteristics

**Section 5.2.5.2 of the CTP**: At screening, the medical examination will include demographics including height and body weight, smoking and alcohol history, relevant medical history and concomitant therapy [...].

Age [years] will be determined as the difference between year of informed consent and year of birth.

BMI will be calculated as weight  $[kg] / (0.01 * height [cm]^2)$ .

#### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

For basic study information on investigational products, assignment of treatment sequences, and selection of doses, please see CTP, Sections 3 and 4.

The study will be performed as a randomised, open-label, two-way crossover trial with 2 treatments (T and R) and 2 treatment sequences (TR or RT).

In total, it was planned to assign 30 healthy male and female subjects to the two treatment sequences in a 1:1 ratio.

For details of dosage and formulation see <u>Table 6.1: 1</u> below:

Table 6.1: 1 Treatments and labels used in the analysis

| Treatment | | Short label | Short label for footnote |
|---|---|---|---|
| T | Empagliflozin 25/Linagliptin 5/<br>Metformin XR 1000 FDC, fed | FDC25 fed | Empa25/Lina5/<br>Met1000 FDC<br>fed |
| R | Empagliflozin 25 + Linagliptin 5 + Metformin XR 2*500, fed | E25+L+M fed | Empa25+Lina5<br>+Met1000 Tab<br>fed |

The following separate study phases will be defined for the analyses of AEs:

- Screening (ranging from 0:00 h on day of informed consent until first administration time of study drug)
- **On treatment** (including residual effect period (REP); i.e. ranging from the time of administration of the respective treatment until 7 days thereafter)
- **Follow-up** (ranging from end of on treatment phase until next drug administration or 0:00 h on the day after trial termination date, according to previous treatment (labelled "FU-Test", "FU-Ref"))

Displays of AEs will be presented separately for the following treatments during on treatment phase:

- Empagliflozin 25/Linagliptin 5/Metformin XR 1000 FDC, fed (labelled "FDC25 fed")
- Empagliflozin 25 + Linagliptin 5 + Metformin XR 2\*500, fed (labelled "E25+L+M fed")

Two types of AE displays will be provided in the report:

A) Section 15.3 and Appendix 16.1.9.2.8 (for ClinicalTrials.gov and EudraCT only) of the CTR displays:

In these displays, the on treatment phase will be analysed (labelled with the name of the study treatment (short label)). Screening and follow-up periods will not be included in this analysis. The following total will be provided in addition (Section 15.3 only):

- a total over all on treatment phases included in this analysis ("Total on treatment")
- B) Section 15.4 and Appendix 16.1.9.2.8 (except for ClinicalTrials.gov and EudraCT) of the CTR displays:
  - Screening
  - On treatment (labelled with the name of the study treatment (short label))
  - Follow-up ("FU-Test" and "FU-Ref")

In Section 16.1.9.2.8 AE tables, the following totals will be provided in addition:

• a total over all study phases ("Total")

Tables of vital signs and laboratory values will present results by the above mentioned on treatment phase.

For detailed information on the handling of the treatments in the O\*C views refer to Technical TSAP ADS plan. In particular, AEs will be counted for test or reference treatment if they occur up to the end of the residual effect period (REP) of 7 days.

#### 6.2 IMPORTANT PROTOCOL VIOLATION

Data discrepancies and deviations from the CTP will be identified for all randomised subjects. Listings of protocol deviations and of unresolved discrepancies will be provided to be discussed at the combined report planning and database lock meeting (RPM/DBLM), e.g. deviations in drug administration, in blood sampling etc. At this meeting, it will be decided whether the discrepant data can be used as they are or whether the data have to be corrected in the clinical database.

Each protocol deviation must be assessed to determine whether it is an important protocol violation. A protocol violation (PV) is important if it affects the rights or safety of the study subjects or if it can potentially influence the primary outcome measure(s) for the respective subjects in a way that is neither negligible nor in accordance with the study objectives. This last category of important PV forms the basis for the decision of whether a subject does or does not belong to an analysis set. PVs that do not influence the subject's rights and safety or the evaluability of the subjects for the main study objectives are called non-important PVs. These are only considered when checking the trial quality in general.

If any important PVs are identified, they are to be summarised into categories and will be captured in the RPM/DBLM minutes via an accompanying Excel spreadsheet [001-MCS-50-413\_RD-02] (2). The following table contains the categories which are considered to be important protocol violations in this trial. If the data show other important PVs, this table will be supplemented accordingly by the time of the RPM/DBLM.

TSAP for BI Trial No: 1361.3 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.2: 1 Important protocol violations

| A Entrance criteria not met A1 Inclusion criteria violated A2 Exclusion criteria violated B Informed consent B1 Informed consent not available B2 Informed consent too late C Trial medication and randomisation C1 Incorrect trial medication taken C2 Randomisation not followed C3 Non-compliance C4 Medication code broken inappropriately C5 Incorrect intake of trial medication C6 Improper washout between treatments D Concomitant medication D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication E Missing data | |
|---|---|
| B Informed consent B1 Informed consent not available B2 Informed consent too late C Trial medication and randomisation C1 Incorrect trial medication taken C2 Randomisation not followed C3 Non-compliance C4 Medication code broken inappropriately C5 Incorrect intake of trial medication C6 Improper washout between treatments D Concomitant medication D1 Prohibited medication not taken D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| B Informed consent B1 Informed consent not available B2 Informed consent too late C Trial medication and randomisation C1 Incorrect trial medication taken C2 Randomisation not followed C3 Non-compliance C4 Medication code broken inappropriately C5 Incorrect intake of trial medication C6 Improper washout between treatments D Concomitant medication D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| B1 Informed consent not available B2 Informed consent too late C Trial medication and randomisation C1 Incorrect trial medication taken C2 Randomisation not followed C3 Non-compliance C4 Medication code broken inappropriately C5 Incorrect intake of trial medication C6 Improper washout between treatments D Concomitant medication D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| B2 Informed consent too late C Trial medication and randomisation C1 Incorrect trial medication taken C2 Randomisation not followed C3 Non-compliance C4 Medication code broken inappropriately C5 Incorrect intake of trial medication C6 Improper washout between treatments D Concomitant medication D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| C Trial medication and randomisation C1 Incorrect trial medication taken C2 Randomisation not followed C3 Non-compliance C4 Medication code broken inappropriately C5 Incorrect intake of trial medication C6 Improper washout between treatments D Concomitant medication D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| C1 Incorrect trial medication taken C2 Randomisation not followed C3 Non-compliance C4 Medication code broken inappropriately C5 Incorrect intake of trial medication C6 Improper washout between treatments D Concomitant medication D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| C2 Randomisation not followed C3 Non-compliance C4 Medication code broken inappropriately C5 Incorrect intake of trial medication C6 Improper washout between treatments D Concomitant medication D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| C3 Non-compliance C4 Medication code broken inappropriately C5 Incorrect intake of trial medication C6 Improper washout between treatments D Concomitant medication D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| C4 Medication code broken inappropriately C5 Incorrect intake of trial medication C6 Improper washout between treatments D Concomitant medication D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| C5 Incorrect intake of trial medication C6 Improper washout between treatments D Concomitant medication D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| C6 Improper washout between treatments D Concomitant medication D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| D Concomitant medication D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| D1 Prohibited medication use D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| D2 Mandatory medication not taken D3 Improper washout of concomitant medication | |
| D3 Improper washout of concomitant medication | |
| E Missing data | |
| E1 Certain violations of procedures used to measure primary or secondary data | |
| F Incorrect timing <sup>1</sup> | |
| F1 Certain violations of time schedule used to measure primary or secondary da | ta |
| G Other trial specific important violations | |
| G1 Incorrect intake of meal | |
| G2 PVs affecting safety and rights | |

Time deviations will only be flagged as important PV, when leading to exclusion of the entire subject from an analysis set Source: 'Protocol Violation Handling Definitions' [001-MCS-50-413\_RD-01] (3)

TSAP for BI Trial No: 1361.3 Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### PATIENT SETS ANALYSED 6.3

Treated set (TS):

This subject set includes all subjects who were documented to have received one dose of study drug.

This is the full analysis set population in the sense of ICH-E9.

It is used for safety analyses.

**Section 7.3.1 of the CTP:** *Plasma concentration data and parameters of a subject will be* included in the statistical pharmacokinetic (PK) analyses if they are not flagged for exclusion due to a protocol violation relevant to the evaluation of PK (to be decided no later than in the Report Planning Meeting) or due to PK non-evaluability (as revealed during data analysis, based on the criteria specified below). Exclusion of a subject's data will be documented in the clinical trial report.

Relevant protocol violations may be:

- Incorrect trial medication taken, that is, the subject received at least one dose of trial medication the subject was not assigned to
- Incorrect dose of trial medication taken
- Use of restricted medications

Plasma concentrations and/or parameters of a subject will be considered as non-evaluable, if for example:

- The subject experiences emesis that occurred at or before 2 times median tmax of the respective treatment (median  $t_{max}$  is to be determined excluding the subjects experiencing emesis)
- A predose concentration is >5%  $C_{max}$  value of that subject
- Missing samples/concentration data at important phases of PK disposition curve
- PK parameter set (PKS):

This subject set includes all subjects in the TS who provide at least one primary or secondary PK parameter that was not excluded according to the description above. Thus, a subject will be included in the PKS, even if he/she contributes only one PK parameter value for one period to the statistical assessment.

The descriptive analysis of PK concentrations will be based on the analysis data set (ADS) ADPC as described at the beginning of Section 7.

Table 6.3: 1 Subject sets analysed

| | Analysis set | |
|------------------------------------------------|--------------|-----|
| Class of endpoint | TS | PKS |
| Analyses of primary and secondary PK endpoints | | X |
| Safety endpoints | X | |
| Demographic/baseline endpoints | X | |
| Important protocol violations | X | |
| Disposition | X | |

#### 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one centre.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Handling of missing data and outliers will be performed as described in the CTP, Section 7.4.

The only exception where imputation might be necessary for safety evaluation are AE dates. Missing or incomplete AE dates are imputed according to BI standards (see 001-MCG-156\_RD-01 (4)).

Missing data and outliers of PK data are handled according to BI standards (see 001-MCS-36-472\_RD-01) (5).

## 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

For vital signs and laboratory parameters the baseline is defined as the measurement at screening.

**Section 6.1 of the CTP:** Exact times of measurements outside the permitted time windows will be documented. The acceptable time windows for screening and end-of-trial examination are given in the CTP Flow Chart.

Study measurements and assessments scheduled to occur 'before' trial medication administration on Day 1 are to be performed and completed within a 3 h-period prior to the trial drug administration.

TSAP for BI Trial No: 1361.3 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Adherence to time windows will be checked via the consistency check listings at the RPM/DBLM.

#### 7. PLANNED ANALYSIS

Safety analysis (refer to Section 7.8) will be performed by and will be presented in Sections 15.1 to 15.4 of the CTR and in Appendix 16.2 and 16.1.9.2.

Inferential statistical analyses of PK endpoints (refer to Section 7.4 and Section 7.5.2) will also be performed by and will be presented in Section 15.5 of the CTR and in Appendix 16.1.9.3.

Descriptive data analysis of PK parameters and concentrations will be performed by BI and presented in Section 15.6 of the CTR.

The format of the listings and tables will follow the standards defined in the BI corporate guideline "Reporting of Clinical Trials and Project Summaries" [001-MCG-159] (6) with the exception of those generated for PK-calculations.

The individual values of all subjects will be listed, sorted by treatment sequence, subject number, visit and actual treatment (if appropriate). The listings will be included in Appendix 16.2 of the CTR.

For end-of-text tables, the set of summary statistics for non-PK parameters is:

N number non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For analyte concentrations as well as for all PK parameters, the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category, as well as the percentage (%) for each treatment group. Percentages will be rounded to one decimal place and will be based on all subjects in the respective subject set whether they have non-missing values or not. The category 'missing' will be displayed only if there are actually missing values.

Units of variables should be given in the titles or column/row descriptors in square brackets (e.g. [mg]).

#### Exclusion of PK parameters

The analysis data set (ADS) ADPP contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS will include parameters if they are not flagged for exclusion, that is APEXCO is equal to "Included".

## Exclusion of PK concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to 'ALL CALC', the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to 'DESC STATS' the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition 'TIME VIOLATION' or 'TIME DEVIATION' the value can be used for further analyses based on actual times. If ACEXCO is set to 'HALF LIFE' the value will be excluded from half-life calculation only; the value is included for all other analyses.

Further details are given in 001-MCS-36-472\_RD-01 "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (5) and 001-MCS-36-472\_RD-03 "Description of Analytical Transfer Files and PK/PD Data Files" (11).

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report, based on the TS.

The data will be summarised by treatment sequence and in total.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Frequency tables are planned for this section of the report, based on the TS.

Concomitant diseases will be coded using the coding system of the Medical Dictionary for Drug Regulatory Activities (MedDRA). Medications will be coded using the World Health Organization Drug Dictionary (WHO-DD). The coding version number will be displayed as a footnote in the respective output.

The diagnoses and medications will be listed. Subjects without any concomitant diagnoses or concomitant therapies should be marked with a "No" in the respective column.

The relevance of the concomitant therapies to the evaluation of PK will be decided no later than at the RPM/DBLM.

#### 7.3 TREATMENT COMPLIANCE

**Section 4.3 of the CTP:** Compliance will be assured by administration of all trial medication in the study centre under supervision of the investigating physician or a designee. The measured plasma concentrations will provide additional confirmation of compliance.

It is not intended to list the compliance separately. Any deviations from complete intake will be addressed in the RPM/DBLM (cf. TSAP <u>Section 6.2</u>) and described in the CTR.

#### 7.4 PRIMARY ENDPOINTS

Bioequivalence is to be determined on the basis of the primary pharmacokinetic endpoints (see Section 5.1).

**Section 7.1.3 of the CTP:** For the bioequivalence analyses, pharmacokinetic endpoints will be log-transformed (natural logarithm) prior to fitting the ANOVA (analysis of variance) model (see below).

## Primary analysis

The statistical model used for the analysis of primary and secondary endpoints will be an ANOVA model on the logarithmic scale. This model will include effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' will be considered as random, whereas the other effects will be considered as fixed. The model is described by the following equation:

$$y_{ijkm} = \mu + \zeta_i + s_{im} + \pi_i + \tau_k + e_{ijkm}$$
, where

 $y_{ijkm} = logarithm \ of \ response \ (endpoint) \ measured \ on \ subject \ m \ in \ sequence \ i \ receiving \ treatment \ k \ in \ period \ j,$ 

 $\mu$  = the overall mean.

$$\zeta_i = the i^{th} sequence effect, i = 1, 2$$

 $s_{im}$  = the effect associated with the  $m^{th}$  subject in the  $i^{th}$  sequence,  $m = 1, 2, ..., n_i$ 

$$\pi_j = the j^{th} period effect, j = 1, 2$$

$$\tau_k = the \ k^{th} \ treatment \ effect, \ k = 1, \ 2$$

 $e_{ijkm}$  = the random error associated with the  $m^{th}$  subject in sequence i who received treatment k in period j.

The following SAS code can be used to fit the model:

```
PROC MIXED DATA=indata;
CLASS subject treatment sequence period;
MODEL logkp = treatment sequence period / DDFM=KR HTYPE=2
SOLUTION CL ALPHA=0.1;
RANDOM subject(sequence) / S;
LSMEANS treatment / PDIFF=CONTROL("Ref_trt") CL ALPHA=0.1;
RUN;
```

The implementation for this analysis will be accomplished by using the XPKISTAT macro, based on PKS, and option BWC (Bioavailability/Bioequivalence, within-subject design, time-controlled).

**Section 7.1.3 of the CTP:** For each endpoint, the difference between the expected means for log(T)-log(R), will be estimated by the difference in the corresponding adjusted means (Least Squares Means), and a two-sided 90% confidence interval (CI) based on the t-distribution will be computed. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% CIs for each endpoint.

#### Further analysis

As a sensitivity analysis, this ANOVA will be repeated for the primary and secondary endpoints with all sources of variation ('sequence', 'subjects within sequences', 'period', 'treatment') considered as fixed effects. This analysis will be done using PROC GLM. The following SAS code can be used to fit the model:

```
PROC GLM DATA=indata;
CLASS subject treatment sequence period;
MODEL logkp = treatment sequence period subject(sequence);
LSMEANS treatment / PDIFF=CONTROL("Ref_trt") CL ALPHA=0.1;
RUN;
```

#### 7.5 SECONDARY ENDPOINTS

## 7.5.1 Key secondary endpoints

This section is not applicable as no key secondary endpoint has been specified in the protocol.

#### 7.5.2 Secondary endpoints

The secondary PK parameter  $AUC_{0-\infty}$  will be assessed using the same methods as described for the primary endpoints but will not be interpreted in a confirmatory sense.

#### 7.7 EXTENT OF EXPOSURE

Descriptive statistics are planned for this section of the report based on the TS. The date and time of drug administration will be listed for each subject.

### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

The safety data for treated subjects who failed to complete the study (dropouts or withdrawals) will be reported as far as their data are available. All withdrawals will be documented and the reason for withdrawal recorded.

#### 7.8.1 Adverse events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature and will be based on BI standards as presented in the corporate guideline: "Analysis and Presentation of Adverse Event Data from Clinical Trials" [001-MCG-156] (8).

The standard AE analyses will be based on the number of subjects with AEs (and not on the number of AEs).

For analysis multiple AE occurrence data on the CRF will be collapsed into an AE provided that all of the following applies:

- All AE attributes are identical (LLT, intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AE of special interest)
- The occurrences were time-overlapping or time-adjacent (time-adjacency of 2 occurrences is given if the second occurrence started within one hour after end of the first occurrence).

For further details on summarization of AE data, please refer to [001-MCG-156] (8,4).

#### **Section 5.2.2.1 of the CTP:** *The following are considered as AESIs in this trial:*

- Hepatic injury, as defined by the following alterations of hepatic laboratory parameters:
  - o an elevation of AST and/or ALT  $\geq$ 3-fold ULN combined with an elevation of total bilirubin  $\geq$ 2-fold ULN measured in the same blood sample, and/or
  - o marked peak aminotransferase (ALT, and/or AST) elevations ≥10 fold ULN

These lab findings constitute a hepatic injury alert and the patients showing these lab abnormalities need to be followed up according to the 'DILI checklist' provided in the ISF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the Investigator should make sure these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

- Pancreatitis
- Hypersensitivity defined as angioedema, severe cutaneous adverse reactions or anaphylactic responses
- Ketoacidosis

The analysis of adverse events will be based on the concept of treatment emergent adverse events.

**Section 5.2.2.2 of the CTP:** The REP for the combined treatment with empagliflozin, linagliptin, and metformin, when measurable drug levels or pharmacodynamic effects are still likely to be present, is defined as 7 days after the last administration of trial medication. Therefore, all AEs which occur through the treatment phase and throughout the REP will be considered as on treatment [...].

All adverse events occurring before first drug administration will be assigned to 'screening', those between intake of trial medication and end of the 7-day REP will be assigned to the corresponding treatment ('on treatment'). AEs occurring after the REP but prior to next drug administration or termination date will be assigned to 'follow-up'. The follow-up will be summarized according to previous treatment.

**Section 7.3.3 of the CTP:** AEs occurring after the last per protocol contact but entered before database lock will be reported to drug safety only and will not be captured in the trial database.

For more detail see the TSAP ADS plan.

According to ICH E3 (9), AEs classified as 'other significant' need to be reported and will include those non-serious and non-significant adverse events with

- (i) 'action taken = discontinuation' or 'action taken = reduced', or
- (ii) marked haematological and other lab abnormalities or lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at the Report Planning Meeting.

An overall summary of AEs (including AESIs) will be presented.

The frequency of subjects with AEs will be summarised by treatment, primary system organ class (SOC) and preferred term (PT). Separate tables will be provided for subjects with other significant AEs according to ICH E3 (9), for subjects with serious AEs, for subjects with drug-related AEs, for subjects with drug related serious adverse events and for subjects with AESIs.

The SOC and PTs will be sorted by frequency. The MedDRA version number will be displayed as a footnote in the respective output.

In addition, frequencies of subjects with non-serious AEs that had an incidence of > 5% for at least one treatment will be summarised by treatment, primary SOC and PT.

For disclosure of adverse events on EudraCT, additional information not included in a standard AE analysis will be performed. The following three entries will be created:

- Adverse Events per arm for disclosure on EudraCT
- Non-serious Adverse Events for disclosure on EudraCT
- Serious Adverse Events for disclosure on EudraCT

#### 7.8.2 Laboratory data

Descriptive statistics will be calculated for screening and end-of-trial visits as well as for the difference from baseline (=screening). The summary statistics will be provided in total. Laboratory data assessed within 7 days prior to the drug administration in the second treatment period will only be listed.

Laboratory data will be analysed qualitatively via comparison of laboratory data to their reference ranges. Values outside the reference range as well as values defined as clinically relevant will be flagged in the data listings.

Frequency tables of changes with respect to the reference range between baseline and last value on treatment will be presented.

Possibly clinically significant abnormal laboratory values are only those identified either in the Investigator's comments on the eCRF or at the RPM/DBLM at the latest. It is the investigator's responsibility to decide whether a lab value is clinically significantly abnormal or not. Standard or project-specific rules for flagging clinically significant values will not be applied in this study.

The analyses of laboratory data will be based on BI standards [001-MCG-157] (10).

#### 7.8.3 Vital signs

Descriptive statistics will be performed for vital signs (blood pressure and pulse rate) for both treatment sequences together (in total).

**Section 7.3.3 of the CTP:** For vital signs the difference from baseline (screening measurements) will be evaluated.

As vital signs are just measured at screening and post examination only these differences from screening will be calculated and presented in a table. In the listing the difference from screening will also be displayed.

Clinically relevant findings in vital signs will be reported as AEs.

#### **7.8.4** ECG

ECG recordings will be checked by the investigator for pathological results. Clinically relevant abnormal findings for ECG will be listed under 'Relevant Medical History / Baseline Conditions' (when they occurred during screening) or will be reported as adverse events (when they occurred during treatment).

## **7.8.5** Others

This section is not applicable as no other variables have been specified in the protocol.

# 8. REFERENCES

1 *CPMP/ICH/363/96*: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version.

9 *CPMP/ICH/137/95*: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version.

TSAP for BI Trial No: 1361.3 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1361.3 

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **10. HISTORY TABLE**

Table 10: 1 History table

| Version | Date | Author | Sections | Brief description of change |
|---|---|---|---|---|
| | (DD-MMM-YY) | | changed | |
| Final | 08-DEC-17 | | None | This is the final TSAP without any |
| | | | | modification |